CLINICAL TRIAL: NCT00208169
Title: Aripiprazole (Abilify) Therapy for Reducing Comorbid Substance Abuse
Brief Title: Abilify Therapy for Reducing Comorbid Substance Abuse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-13685
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-08-24 (Estimated); Status verified 2007-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depressive Disorder; Anxiety Disorders; Substance Abuse
Keywords: Comorbid substance abuse/dependence; Comorbid diagnoses; Substance abuse and/or dependence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Anxiety Disorders; Substance-Related Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Aripiprazole start dose at 5 mg/day by day 4-6 increase to 10 mg/da and day 7 and subsequent visits flexible dosing from 10 up to 30 mg/day.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
It is hypothesized that the use of aripiprazole (Abilify) in patients with alcohol and/or drug dependence with comorbid psychiatric conditions will lead to:

* Reduction in the amount of alcohol and/or drugs used as measured by the Time Line Follow Back (TLFB) and the Addiction Severity Index (ASI)
* Reduction in cravings for alcohol and drugs as measured by the Penn Alcohol Craving Scale
* Reduction in symptoms of co-morbid psychiatric disorders compared to before starting aripiprazole.

DETAILED DESCRIPTION:
Substance abuse disorders are a major public health problem. With a current prevalence rate of 18%, substance abuse and dependence costs the nation over $300 billion per year in treatment costs and lost productivity. Approximately 20% of all patients attending primary care clinics and 35% of all patients attending psychiatric clinics meet Diagnostic and Statistical Manual IV (DSM IV) criteria for substance abuse or dependence.

The treatment of substance abuse and dependence disorders is complex and involves individual and group therapy, maintenance of sobriety, commitment to structured living, and participation in self-help groups. To date, pharmacotherapy for substance dependence disorders has had limited success. Several medications have been tested in the past, including tricyclic antidepressants, selective serotonin reuptake inhibitors, buspirone, bupropion, venlafaxine, nefazodone, bromocriptine, amantadine, naltrexone, and acamprosate. Of these, naltrexone has obtained an FDA indication for treatment of alcohol dependence, and acamprosate is in use in Europe. However, these medications are effective in only a relatively small proportion of patients. Benzodiazepines may be useful in treatment of withdrawal syndromes, but their potential for abuse and dependence limits their use in maintenance treatment.

This is an open label pilot study of aripiprazole therapy in the treatment of patients with substance use disorders and co-morbid disorders like Schizophrenia, Schizoaffective disorder, Bipolar disorder, Major depressive disorder, Anxiety (Panic disorder, Generalized Anxiety Disorder, Post-Traumatic Stress Disorder). While Aripiprazole has been approved for the treatment of Schizophrenia, its use in other psychiatric disorders is off label use. Increasing evidence suggests that Aripiprazole might offer some benefit for other psychiatric disorders besides Schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 19 - 65
2. Diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, or anxiety (panic disorder, generalized anxiety disorder, or post-traumatic stress disorder) as confirmed by Mini International Neuropsychiatric Interview (MINI) structured assessment
3. Diagnosis of comorbid substance abuse/dependence as confirmed by the MINI structured assessment
4. Ability to provide signed informed consent
5. Stable general medical health
6. Ability to attend outpatient research clinic.

Exclusion Criteria:

1. Dangerous to self or others
2. Pregnancy, or inability or unwillingness to use approved methods of birth control
3. Inability or unwillingness to provide signed informed consent
4. Inability to attend outpatient research clinic
5. Medical conditions, which would preclude use of aripiprazole
6. Absolute need for ongoing treatment with antipsychotic other than aripiprazole
7. Medical instability defined as likelihood of needing to change prescription medication during the course of the study
8. Patients with prior unsuccessful treatment with aripiprazole
9. Patients with a psychiatric diagnosis of only antisocial personality disorder or only an eating disorder and comorbid substance abuse/dependence.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be days of abstinence during the 12-week follow-up, as measured by the Time Line Follow Back Scale (TLFBS) and the Addiction Severity Index (ASI). | Two years

SECONDARY OUTCOMES:
Secondary outcome measures will assess severity of symptoms as measured by the Hamilton Depression Rating Scale (HAM-D), Hamilton Anxiety Scale (HAM-A), Young Mania Rating Scale (YMRS), and the Brief Psychiatric Rating Scale (BPRS) | Two years
The Penn Alcohol Craving Scale will also be used. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Pirzada S. Sattar, M.D., Principal Investigator — Creighton University
Locations (1):
- Creighton University Psychiatry and Research Center, Omaha, Nebraska, United States